CLINICAL TRIAL: NCT02069535
Title: An Open Trial to Assess the Tolerability of AVANZ® Cupressus Immunotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-X-03; 2013-004720-11 (EudraCT Number)
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Cupressus arizonica

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AVANZ Cupressus (Experimental): AVANZ Cupressus
  Interventions: Biological: AVANZ Cupressus

INTERVENTIONS:
Biological: AVANZ Cupressus — AVANZ Cupressus

SUMMARY:
This trial is an open, national, multi-centre trial. The main objective of this trial is to assess the tolerability of the up-dosing phase of AVANZ® Cupressus arizonica by measurement of related Adverse Events.

DETAILED DESCRIPTION:
The main objective of this trial is to assess the tolerability of the up-dosing phase of AVANZ® Cupressus arizonica, the measurement rate is the frequency of patients with investigational medicinal product (IMP)-related adverse events (AEs) will be the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* A documented clinically relevant history of Cupressus arizonica pollen induced allergic rhinoconjunctivitis with or without asthma for at least one year prior to trial entry.
* Positive Skin Prick Test (SPT) response to Cupressus arizonica pollen (wheal diameter ≥ 3 mm)

Exclusion Criteria:

* History of severe asthma exacerbation or emergency room visit or admission for asthma in the previous 12 months.
* Previous treatment with immunotherapy with Cupressus arizonica pollen extract within the last 5 years (initiation of subcutaneous immunotherapy is acceptable if treatment has been discontinued before reaching maintenance dose; for SLIT 3 months in the last 5 years is accepted).
* Ongoing treatment with any allergen-specific immunotherapy product.
* A history of anaphylaxis with cardiorespiratory symptoms (immunotherapy, exercise-induced, food allergy, drugs or an idiopathic reaction).
* A systemic disease affecting the immune system (e.g. insulin-dependent diabetes, autoimmune disease, immune complex disease, or immune deficiency disease whether acquired or not).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Frequency of patients with IMP-related AEs | 6 treatment weeks

SECONDARY OUTCOMES:
Frequency of patients with systemic reactions | 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Fernández Rivas, PhD, Study Chair — Hospital Clínico Universitario San Carlos, Madrid
Locations (1):
- Hospital Clinico Universitario San Carlos, Madrid, Madrid, Spain